CLINICAL TRIAL: NCT03132259
Title: Comparative Low and High Dose of Dexmedethomidine Can Stabilize Hemodynamics and Blood Loss in Pituitary Tumor Removal by Transphenoid Approach
Brief Title: Comparative Low and High Dose of Dexmedethomidine in Pituitary Tumor Removal by Transphenoid Approach
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, SMuangman, Assisted Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116/2559
Record Dates: First submitted 2016-07-18; First posted 2017-04-27 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Pituitary Tumor
Keywords: Dexmedethomidine
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose dexmedethomidine (Experimental): High dose is 0.5 microgram/kg/hr
  Interventions: Drug: high dose dexmedethomidine
- Low dose dexmedethomidine (Experimental): Low dose is 0.2 microgram/kg/hr
  Interventions: Drug: low dose dexmedethomidine

INTERVENTIONS:
Drug: high dose dexmedethomidine — Dexmedethomidine continuous drip 0.5 mcg/kg/hr a
  Other Names: Precedex
  Arms: High dose dexmedethomidine
Drug: low dose dexmedethomidine — Dexmedethomidine continuous drip 0.2 mcg/kg/hr
  Arms: Low dose dexmedethomidine

SUMMARY:
Transnasal transsphenoidal (TNTS) resection of pituitary tumors involves wide fluctuation in hemodynamic parameter and causes hypertension and tachycardia due to intense noxious stimuli during various stages of surgery. None of routinely used anesthetic agents effectively blunts the undesirable hemodynamic responses, and therefore usually there is a need to use increased doses of anesthetic agents. Dexmedetomidine (DEX) an α-2 adrenergic receptor agonist, because its sympatholytic and antinociceptive properties may ensure optimal intraoperative hemodynamic stability during critical moments of surgical manipulation. In addition, DEX reduced the anesthetic requirement with rapid recovery at the end of surgery. The main aim of the study was to evaluate the effect of DEX on perioperative hemodynamics, anesthetic requirements

DETAILED DESCRIPTION:
DEX as an anesthetic adjuvant improved hemodynamic stability and decreased anesthetic requirements in patients undergoing TNTS resection of pituitary tumor. In addition, DEX provided better surgical field exposure conditions and early recovery from anesthesia

ELIGIBILITY:
Inclusion Criteria:

1. Age18-65
2. ASA 1-2
3. Elective TNTS resection of Pituitary Tumor
4. No narcotic before surgery as premedication
5. Able to Extubate

Exclusion Criteria:

1. GCS less than 15
2. Preoperative Heart Rate less than 50 beat/min
3. No Beta-Blockers
4. Pregnant patients
5. Take any Alpha-Methyldopa, Clonodine, Other Alpha-2 Adrenergic Agonist
6. Hemodynamic unstable
7. Systolic BP more than 160mmHg
8. CAD
9. Renal insuffuciency
10. Allergy in dexmedethomidine and opioid
11. BMI more than 30
12. Denied consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Comparative Low and High Dose of Dexmedethomidine in Pituitary Tumor Removal by Transphenoid Approach | 24 hours
  Low dose is 0.2microgram/kg/hr High dose is 0.5 microgram/kg/hr what is the dose proper and hemodynamic changes. Hemodynamic change means BP is lower than 20% of baseline more than 10minute

SECONDARY OUTCOMES:
Comparative Low and High Dose of Dexmedethomidine in Pituitary Tumor | 24 hours
  Low dose is 0.2microgram/kg/hr High dose is 0.5 microgram/kg/hr how much dose blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Saipin Muangman, physician, Principal Investigator — Mahidol University
Locations (1):
- Faculy of Medicine Siriraj hospital Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gopalakrishna KN, Dash PK, Chatterjee N, Easwer HV, Ganesamoorthi A. Dexmedetomidine as an Anesthetic Adjuvant in Patients Undergoing Transsphenoidal Resection of Pituitary Tumor. J Neurosurg Anesthesiol. 2015 Jul;27(3):209-15. doi: 10.1097/ANA.0000000000000144. PMID 25493927
- [Result] Anjum N, Tabish H, Debdas S, Bani HP, Rajat C, Anjana Basu GD. Effects of dexmedetomidine and clonidine as propofol adjuvants on intra-operative hemodynamics and recovery profiles in patients undergoing laparoscopic cholecystectomy: A prospective randomized comparative study. Avicenna J Med. 2015 Jul-Sep;5(3):67-73. doi: 10.4103/2231-0770.160231. PMID 26229757
- [Result] Polat R, Peker K, Baran I, Bumin Aydin G, Topcu Guloksuz C, Donmez A. Comparison between dexmedetomidine and remifentanil infusion in emergence agitation during recovery after nasal surgery: A randomized double-blind trial. Anaesthesist. 2015 Oct;64(10):740-6. doi: 10.1007/s00101-015-0077-8. Epub 2015 Sep 2. PMID 26329913
- [Result] Karwacki Z, Niewiadomski S, Rzaska M, Witkowska M. The effect of bispectral index monitoring on anaesthetic requirements in target-controlled infusion for lumbar microdiscectomy. Anaesthesiol Intensive Ther. 2014 Sep-Oct;46(4):284-8. doi: 10.5603/AIT.2014.0046. PMID 25293480